CLINICAL TRIAL: NCT01843374
Title: A Phase 2b, Randomized, Double-blind Study Comparing Tremelimumab to Placebo in Second- or Third-line Treatment of Subjects With Unresectable Pleural or Peritoneal Malignant Mesothelioma
Brief Title: Randomized, Double-blind Study Comparing Tremelimumab to Placebo in Subjects With Unresectable Malignant Mesothelioma
Acronym: Tremelimumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4880C00003; 2012-003524-21 (EudraCT Number)
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Unresectable Pleural or Peritoneal Malignant Mesothelioma
Keywords: tremelimumab; pleural, peritoneal; malignant mesothelioma; CTLA-4
MeSH Terms: conditions — Mesothelioma, Malignant; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — tremelimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tremelimumab (Experimental): Tremelimumab
  Interventions: Drug: Tremelimumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab is to be administered as an IV solution, followed by observation.
  Arms: Tremelimumab
Drug: Placebo — Placebo is to be administered as an IV solution, followed by observation.
  Arms: Placebo

SUMMARY:
This is a Phase 2b, randomized, double-blind, parallel-group study. Subjects with unresectable pleural or peritoneal malignant mesothelioma will be randomized in a 2:1 ratio to receive either tremelimumab or placebo. Approximately 564 subjects will be enrolled at study centers in multiple countries. The study consists of a screening period, a treatment period, a 90-day follow-up period for safety, and a long-term survival follow-up period.

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, parallel-group study. Subjects with unresectable pleural or peritoneal malignant mesothelioma will be randomized in a 2:1 ratio to receive either tremelimumab or placebo.

Randomization will be stratified by EORTC status (low-risk vs high-risk), line of therapy (second vs third), and anatomical site (pleural vs peritoneal). This study plans to use the EORTC to stratify subjects into high or low risk groups in order to ensure balanced randomization to the different treatment groups. For subjects in whom pemetrexed was contraindicated or not tolerated or not an approved therapy (eg, peritoneal mesothelioma), prior therapy with a first-line platinum-based regimen is required. Approximately 564 subjects will be enrolled at study centers in multiple countries.

The study consists of a screening period, a treatment period, a 90-day follow-up period for safety, and a long-term survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed pleural or peritoneal malignant mesothelioma;
2. Disease not amenable to curative surgery;
3. Age 18 and over at the time of consent;
4. ECOG Performance status 0-1;
5. Progressed after previous receipt of 1-2 prior systemic treatments for advanced disease that included a first-line pemetrexed (or anti-folate)-based regimen in combination with platinum agent.
6. Recovered from all toxicities associated with prior treatment, to acceptable baseline status, or a NCI CTCAE Grade of 0 or 1, except for toxicities not considered a safety risk,
7. Measurable diseaseby modified RECIST for pleural mesothelioma or RECIST v1.1 for peritoneal mesothelioma;
8. Adequate bone marrow, hepatic, and renal function determined within 14 days prior to randomization defined as:
9. Negative screening test results for human immunodeficiency virus (HIV), hepatitis A, B and C.
10. Written informed consent and any locally required authorization (eg, HIPAA in the USA, EU Data Privacy Directive authorization in the EU) obtained from the subject/legal representative prior to performing any protocol- related procedures, including screening evaluations;
11. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician.
12. Nonsterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Days 1 through 90 post last dose. In addition, they must refrain from sperm donation for 90 days after the final dose of investigational product.

Exclusion Criteria:

1. Subjects who failed more than 2 prior systemic treatment regimens for advanced malignant mesothelioma;
2. Received any prior mAb against CTLA-4, programmed cell death 1 (PD1) or programmed cell death 1 ligand 1 (PD-L1);
3. History of chronic inflammatory or autoimmune disease with symptomatic disease within the last 3 years prior to randomization.
4. Active, untreated central nervous system (CNS) metastasis
5. Any serious uncontrolled medical disorder or active infection that would impair the subject's ability to receive investigational product;
6. History of other malignancy unless the subject has been disease-free for at least 3 years;
7. Pregnant or breast feeding at time of consent;
8. Any condition that would prohibit the understanding or rendering of information and consent and compliance with the requirements of this protocol;
9. Active or history of diverticulitis;
10. Active or history of inflammatory bowel disease, irritable bowel disease, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea. Active or history of systemic lupus erythematosus or granulomatosis with polyangiitis;
11. History of sarcoidosis syndrome;
12. Currently receiving systemic corticosteroids or other immunosuppressive medications or has a medical condition that requires the chronic use of corticosteroids.
13. Subjects should not be vaccinated with live attenuated vaccines within one month prior to starting tremelimumab treatment;
14. The last dose of prior chemotherapy or radiation therapy was received less than 2 weeks prior to randomization;
15. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of vitiligo and alopecia;
16. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results;
17. Concurrent enrollment in another clinical study or receipt of an investigational product within the last 4 weeks
18. Employees of the study site directly involved with the conduct of the study, or immediate family members of any such individuals;
19. Subjects with a history of hypersensitivity to compounds of similar biologic composition to tremelimumab or any constituent of the product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2016-01-24 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (99):
- United States (20):
  - Research Site, Scottsdale, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Durham, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Australia (10):
  - Research Site, Adelaide
  - Research Site, Auchenflower
  - Research Site, Box Hill
  - Research Site, Chermside
  - Research Site, East Bentleigh
  - Research Site, Gosford
  - Research Site, Heidelberg
  - Research Site, Nedlands
  - Research Site, Saint Leonards
  - Research Site, Waratah
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Sainte-Foy, Quebec
- Research Site, Copenhagen, Denmark
- France (7):
  - Research Site, Caen
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Rennes
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (10):
  - Research Site, Berlin
  - Research Site, Esslingen a.N.
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hemer
  - Research Site, Karlsruhe
  - Research Site, Löwenstein
  - Research Site, Lübeck
- Hungary (2):
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Törökbálint
- Research Site, Beersheba, Israel
- Italy (12):
  - Research Site, Alessandria
  - Research Site, Aviano
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Candiolo
  - Research Site, Genova
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Rozzano
  - Research Site, Siena
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Rotterdam
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Research Site, Craiova, Romania
- Russia (3):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
- South Africa (2):
  - Research Site, Kraaifontein
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Jeonnam
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Madrid
  - Research Site, Sabadell (Barcelona)
  - Research Site, Seville
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Umeå
- United Kingdom (8):
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Plymouth
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Baverel P, Roskos L, Tatipalli M, Lee N, Stockman P, Taboada M, Vicini P, Horgan K, Narwal R. Exposure-Response Analysis of Overall Survival for Tremelimumab in Unresectable Malignant Mesothelioma: The Confounding Effect of Disease Status. Clin Transl Sci. 2019 Sep;12(5):450-458. doi: 10.1111/cts.12633. Epub 2019 Apr 12. PMID 30883000
- [Derived] Maio M, Scherpereel A, Calabro L, Aerts J, Perez SC, Bearz A, Nackaerts K, Fennell DA, Kowalski D, Tsao AS, Taylor P, Grosso F, Antonia SJ, Nowak AK, Taboada M, Puglisi M, Stockman PK, Kindler HL. Tremelimumab as second-line or third-line treatment in relapsed malignant mesothelioma (DETERMINE): a multicentre, international, randomised, double-blind, placebo-controlled phase 2b trial. Lancet Oncol. 2017 Sep;18(9):1261-1273. doi: 10.1016/S1470-2045(17)30446-1. Epub 2017 Jul 17. PMID 28729154
- See also: FINAL Redacted PROTOCOL_ 03Jan2017 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=180&filename=FINAL%20Redacted%20PROTOCOL_%2003Jan2017.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 658 patients were screened, 87 patients were excluded from randomisation and 571 patients were randomised:
  Of the 78 excluded, 66 did not meet inclusion/exclusion criteria; 19 withdrew consent and 2 were excluded for other reasons.
Groups:
- TREMELIMUMAB: TREMELIMUMAB 10 mg/kg
Period: Overall Study
Arm/Group | PLACEBO | TREMELIMUMAB
Started | 189 | 382
RANDOMIZED | 189 | 382
Completed | 0 | 3
Not Completed | 189 | 379
Not completed — Death | 155 | 313
Not completed — Withdrawal by Subject | 14 | 20
Not completed — Withdrawing due to Other reason | 20 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TREMELIMUMAB | PLACEBO | Total
Number analyzed (Participants) | 382 | 189 | 571
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (9.24) | 66.3 (8.8) | 65.6 (9.10)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 162 | 75 | 237
  >= 65 years | 220 | 114 | 334
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 38 | 137
  Male | 283 | 151 | 434

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) by treatment arm
Time Frame: 3 years.
Population: ITT population
Measure: Number; unit: Number of Participants
Units Other Than Participants: Participants
Arm/Group | PLACEBO | TREMELIMUMAB
Number analyzed (Participants) | 189 | 382
Number analyzed (Participants) | 189 | 282
Number of Participants
  Number of patients with Events (Death) | 154 | 307
  Number patients censored <= 2 weeks before DCO | 25 | 58
  Number of patients censored > 2 weeks before DCO | 10 | 17
Statistical Analysis 1: Comparison: PLACEBO vs TREMELIMUMAB; H0: No difference between tremelimumab and placebo H1: Difference between tremelimumab and placebo; Test type: Superiority or Other; p = 0.4081, Log Rank — P-value was estimated using the method of Klein et al. 2007 and Whitehead and Whitehead 1991, stratified by EORTC status and Line of therapy; The stratification factors included EORTC status and line of therapy as recorded in IVRS/IWRS; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.76 to 1.12] — Tremelimumab represents the numerator and Placebo the denominator

2. Secondary Outcome: OS Rate at 18 Months by Treatment Arm
Description: The percentage of patients still alive at 18 months
Time Frame: 18 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Units Other Than Participants: Participants
Groups:
- TREMELIMUMAB: Tremelimumab 10mg/kg
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 382 | 189
Percentage of Participants | 17.4 [13.4 to 21.8] | 18.2 [12.7 to 24.5]
Statistical Analysis 1: Comparison: TREMELIMUMAB vs PLACEBO; Test type: Superiority or Other; p = 0.926, Log Rank — Estimated using the methods of Klein et al. 2007 and Whitehead and Whitehead 1991, stratified by EORTC status and line of therapy; Hazard Ratio (HR) = 1.011, 95% CI 2-sided [0.793 to 1.289] — Tremelimumab is the numerator and Placebo the denominator

3. Secondary Outcome: Progression-free Survival by Treatment Arm
Description: Progression-free survival will be measured from randomization to the first documentation of disease progression or death due to any cause, whichever occurs first. Progression is defined using the modified Response Evaluation Criteria in Solid Tumours (RECIST) for pleural mesothelioma or RECIST v1.1 for peritoneal mesothelioma and assessed by computed tomography (CT) or magnetic resonance imaging (MRI), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from randomization to disease progression or death, whichever occurs first, assessed up to 3 years.
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Units Other Than Participants: Participants
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 382 | 189
Months | 2.69 [2.66 to 2.76] | 2.76 [2.76 to 2.79]
Statistical Analysis 1: Comparison: TREMELIMUMAB vs PLACEBO; Test type: Superiority or Other; p = 0.0325, Log Rank — [p-value comment as in outcome 2, analysis 1]; Stratification factors were EORTC status and Line of therapy; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.68 to 0.98] — Tremelimumab is the numerator and placebo, the denominator

4. Secondary Outcome: Overall Response Rate by Treatment Arm
Description: Overall response rate is defined as the proportion of participants with confirmed CR or PR per the modified Response Evaluation Criteria in Solid Tumours (RECIST) for pleural mesothelioma or RECIST v1.1 for peritoneal mesothelioma and assessed by computed tomography (CT) or magnetic resonance imaging (MRI). Complete Response (CR) corresponds to disappearance of all target lesions, and Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) = CR + PR.
Time Frame: Time from randomization to best response to treatment, assessed up to 3 years.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage
Units Other Than Participants: Participants
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 382 | 189
Percentage | 4.5 [2.6 to 7.0] | 1.1 [0.1 to 3.8]

5. Secondary Outcome: Duration of Response by Treatment Arm
Description: Duration of response will be defined as the duration from the first documentation of complete response (CR), partial response (PR) to the first documented disease progression.
Time Frame: Duration of response from the first documentation of objcetive response (confirmed CR or PR) to the first documented disease progression, assessed up to 14 weeks after the initial response.
Population: ITT
Measure: Median (Full Range); unit: Months
Units Other Than Participants: Participants
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 382 | 189
Months | 4.8 [0 to 13.4] | 5.57 [2.8 to 8.3]

6. Secondary Outcome: Disease Control Rate by Treatment Arm
Description: Disease control rate (DCR) is defined as the proportion of participants with best response of complete response (CR), partial response (PR), or stable disease (SD) of ≥ 12 weeks duration
Time Frame: Time from randomization to disease progression or death, whichever occurs first, assessed up to 3 years.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage
Units Other Than Participants: Participants
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 382 | 189
Percentage | 21.7 [16.0 to 28.3] | 27.7 [23.3 to 32.5]

7. Secondary Outcome: Durable Disease Control Rate by Treatment Arm
Description: Durable disease control rate (DDCR) is defined as the percentage of participants with best response of complete response (CR), partial response (PR), or stable disease (SD) of ≥ 6 months duration
Time Frame: Time from randomization to disease progression or death, whichever occurs first, assessed up to 3 years.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage
Units Other Than Participants: Participants
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 382 | 189
Percentage | 16.8 [13.1 to 20.9] | 11.6 [7.4 to 17.1]

8. Secondary Outcome: Number of Participants Reporting Any Adverse Event
Description: Any untoward medical occurrence in a patient or clinical investigation participants administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Day 1- 90 days post dose
Population: Safety population
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | TREMELIMUMAB | PLACEBO
Number analyzed (Participants) | 380 | 189
Participants | 364 | 179

9. Secondary Outcome: Number of Participants Reporting Any Serious Adverse Events
Time Frame: Day 1 to 90 days post dose
Population: Safety population
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | PLACEBO | TREMELIMUMAB
Number analyzed (Participants) | 189 | 380
Participants | 85 | 218

10. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies
Description: The immunogenicity titer is reported for samples confirmed positive for the presence of anti tremelimumab antibodies.
Time Frame: Week 5
Population: Safety population
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | PLACEBO | TREMELIMUMAB
Number analyzed (Participants) | 188 | 377
Participants | 0 | 15

ADVERSE EVENTS:
Arm/Group | PLACEBO | TREMELIMUMAB
All-Cause Mortality (participants affected / at risk) | 160/189 | 318/382
Serious Adverse Events (participants affected / at risk) | 85/189 | 218/380
Other Adverse Events (participants affected / at risk) | 159/189 | 338/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=189) | TREMELIMUMAB (N=380)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (7)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (4)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (4)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (2)
Pericardial effusion (Cardiac disorders) | 6 (6) | 9 (10)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Hypophysitis (Endocrine disorders) | 0 (0) | 3 (3)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Lymphocytic hypophysitis (Endocrine disorders) | 0 (0) | 3 (3)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (10) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 24 (27)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 69 (106)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 9 (11)
Oesophageal compression (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 5 (5)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (9) | 12 (13)
Asthenia (General disorders) | 3 (3) | 4 (5)
Device breakage (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (2)
Early satiety (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (4)
General physical health deterioration (General disorders) | 4 (4) | 9 (10)
Malaise (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 2 (2)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 11 (12)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (3)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Lung infection (Infections and infestations) | 2 (2) | 5 (8)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (8) | 11 (13)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 6 (7)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 10 (12)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (2)
Syncope (Nervous system disorders) | 3 (4) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 5 (5)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (31) | 29 (33)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Social problem (Social circumstances) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Inferior vena cava stenosis (Vascular disorders) | 1 (1) | 0 (0)
Inferior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=189) | TREMELIMUMAB (N=380)
Anaemia (Blood and lymphatic system disorders) | 23 (37) | 54 (76)
Abdominal distension (Gastrointestinal disorders) | 13 (14) | 16 (18)
Abdominal pain (Gastrointestinal disorders) | 22 (31) | 44 (54)
Constipation (Gastrointestinal disorders) | 53 (62) | 65 (82)
Diarrhoea (Gastrointestinal disorders) | 35 (49) | 168 (368)
Nausea (Gastrointestinal disorders) | 38 (50) | 103 (126)
Vomiting (Gastrointestinal disorders) | 16 (17) | 71 (91)
Asthenia (General disorders) | 24 (28) | 52 (75)
Fatigue (General disorders) | 60 (72) | 91 (119)
Non-cardiac chest pain (General disorders) | 10 (13) | 17 (21)
Oedema peripheral (General disorders) | 16 (16) | 39 (45)
Pyrexia (General disorders) | 16 (18) | 53 (81)
Urinary tract infection (Infections and infestations) | 4 (5) | 21 (24)
Weight decreased (Investigations) | 17 (18) | 47 (54)
Decreased appetite (Metabolism and nutrition disorders) | 45 (52) | 110 (139)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 21 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 25 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 21 (24)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 33 (41) | 47 (64)
Headache (Nervous system disorders) | 6 (8) | 20 (23)
Anxiety (Psychiatric disorders) | 13 (13) | 20 (20)
Insomnia (Psychiatric disorders) | 13 (13) | 29 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 66 (83)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 60 (79) | 103 (127)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 17 (18)
Night sweats (Skin and subcutaneous tissue disorders) | 10 (10) | 13 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (19) | 103 (157)
Rash (Skin and subcutaneous tissue disorders) | 14 (16) | 76 (113)

LIMITATIONS AND CAVEATS:
Baseline characteristics and efficacy outcomes are from the primary analysis reported in the main CSR based on a DCO of 24th January 2016. Participant flow and AE results are from the CSR Addendum based on a DBL of 23 January 2017.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the communication of results, it being understood that results shall be published regardless of outcome